CLINICAL TRIAL: NCT04110379
Title: Effect of Virtual Reality Glasses as a Distraction Method on Child's Anxiety During Dental Treatment(Randomized Controlled Clinical Trial)
Brief Title: Effect of Virtual Reality Glasses as a Distraction Method on Child's Anxiety During Dental Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Instructor of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VR for anxiety
Record Dates: First submitted 2019-09-24; First posted 2019-10-01 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Dental Anxiety
Keywords: virtual reality; distraction; salivary cortisol

STUDY DESIGN:
Intervention Model Description: The eligible participants will be randomly and equally divided into group I (study) and group II (control). Each group will be further subdivided according to age into subgroup A (preschool aged children) and subgroup B (school aged children).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (VR) (Experimental): Child behavior management will be done using virtual reality glasses distraction (Remax Fantasy Land virtual reality glasses (Schenzen Remax Co.,Ltd))
  Interventions: Behavioral: Virtual Reality (VR)
- Conventional Behavior Management (Active Comparator): Child behavior management will be done using conventional behavior management techniques
  Interventions: Behavioral: Conventional Behavior Management Techniques

INTERVENTIONS:
Behavioral: Virtual Reality (VR) — All the dental procedures that will be done will be explained to the child using tell-show-do technique. VR glasses will be introduced to the child using tell-show-do technique and he will be given a choice of cartoon episodes to select from according to his own interest and age appropriate to view during the dental treatment. The child will be given five minutes to get familiar with the VR glasses before starting the dental treatment.
  Arms: Virtual Reality (VR)
Behavioral: Conventional Behavior Management Techniques — Conventional behavior management techniques will be done to relieve the child's dental anxiety during the dental treatment such as : tell-show-do technique, distraction, and positive reinforcement, according to the child's behavior.
  Arms: Conventional Behavior Management

SUMMARY:
The aim of the study is to evaluate and compare the effect of virtual reality glasses (VR) to conventional behavior management techniques as a distraction method on child's dental anxiety during dental treatment

DETAILED DESCRIPTION:
The study to be conducted will be a randomized controlled clinical trial .The sample will consist of forty children presented to the Department of Pediatric Dentistry and Dental Public Health, 20 preschoolers of age ranging from 4-5 years old and 20 schoolers of age ranging from 6-8 years old. The eligible participants will be randomly divided into a study group where virtual reality glasses distraction will be used for child behavior management and a control group where conventional behavior management techniques (tell-show-do, distraction, and positive reinforcement) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children (ASA category I).
* Frankl behavior rating score 2 or 3.
* Requiring pulpotomy in one of their primary molars.

Exclusion Criteria:

* Children taking medications that interfere with measures of salivary cortisol.
* Presence of any systemic or mental disease.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

PRIMARY OUTCOMES:
Preoperative Venham clinical anxiety rating scale | Baseline; at the beginning of the visit
  This scale consists of 6 categories (range from 0 to 5) where 0= relaxed, 1=uneasy, 2= tense, 3= reluctant, 4= interference, 5= out of contact
Postoperative Venham clinical anxiety rating scale | post dental treatment; after 2 hours
  This scale consists of 6 categories (range from 0 to 5) where 0= relaxed, 1=uneasy, 2= tense, 3= reluctant, 4= interference, 5= out of contact
Preoperative evaluation of salivary cortisol level | Baseline; at the beginning of the visit
  Each child will be asked to pool saliva in his/her mouth for 5 minutes and then passively drool it in the receiving vessel. The whole unstimulated salivary samples obtained will be centrifuged and 2 ml of each sample will be stored at -20º until being processed. The salivary samples will be analyzed for salivary cortisol using solid phase enzyme linked immunosorbent assay using DRG salivary cortisol ELISA kit.
Postoperative evaluation of salivary cortisol level | post dental treatment; after 2 hours
  Each child will be asked to pool saliva in his/her mouth for 5 minutes and then passively drool it in the receiving vessel. The whole unstimulated salivary samples obtained will be centrifuged and 2 ml of each sample will be stored at -20º until being processed. The salivary samples will be analyzed for salivary cortisol using solid phase enzyme linked immunosorbent assay using DRG salivary cortisol ELISA kit.

CONTACTS AND LOCATIONS:
Overall Officials: Yomna Alaa Eldin, BDS, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Karin M.L. Dowidar, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt; Laila El Habashy, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt; Akram Deghady, PhD, Study Director — Faculty of Medicine, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Al-Khotani A, Bello LA, Christidis N. Effects of audiovisual distraction on children's behaviour during dental treatment: a randomized controlled clinical trial. Acta Odontol Scand. 2016 Aug;74(6):494-501. doi: 10.1080/00016357.2016.1206211. Epub 2016 Jul 13. PMID 27409593
- [Background] Appukuttan DP. Strategies to manage patients with dental anxiety and dental phobia: literature review. Clin Cosmet Investig Dent. 2016 Mar 10;8:35-50. doi: 10.2147/CCIDE.S63626. eCollection 2016. PMID 27022303
- [Background] Asl Aminabadi N, Erfanparast L, Sohrabi A, Ghertasi Oskouei S, Naghili A. The Impact of Virtual Reality Distraction on Pain and Anxiety during Dental Treatment in 4-6 Year-Old Children: a Randomized Controlled Clinical Trial. J Dent Res Dent Clin Dent Prospects. 2012 Fall;6(4):117-24. doi: 10.5681/joddd.2012.025. Epub 2012 Nov 12. PMID 23277857
- [Background] Fakhruddin KS, Hisham EB, Gorduysus MO. Effectiveness of audiovisual distraction eyewear and computerized delivery of anesthesia during pulp therapy of primary molars in phobic child patients. Eur J Dent. 2015 Oct-Dec;9(4):470-475. doi: 10.4103/1305-7456.172637. PMID 26929683
- [Background] Gadicherla S, Shenoy RP, Patel B, Ray M, Naik B, Pentapati KC. Estimation of salivary cortisol among subjects undergoing dental extraction. J Clin Exp Dent. 2018 Feb 1;10(2):e116-e119. doi: 10.4317/jced.54369. eCollection 2018 Feb. PMID 29670727